CLINICAL TRIAL: NCT06775496
Title: Life-threatening Infection in Humans: from Epidemiological Analysis to Molecular Genetics
Acronym: QUI_IMMUNO
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: QUI_IMMUNO
Record Dates: First submitted 2024-12-03; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-09

CONDITIONS: Life-threatening Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study, aims to identify and calculate the prevalence of cases potentially associated with congenital errors of immunity (ECI) among patients, hospitalized with infectious disease and carry out their clinical-laboratory characterization. Diagnoses of ECI are becoming increasingly common, by virtue of the continuing discoveries of new disease-causing genes and an increasing understanding of the clinical signs and symptoms of these entities.

The most important challenge still remains to achieve early diagnosis, which is essential for appropriate and individualized treatment that also takes into account the prognostic and genetic counseling aspect related to these disorders, which are associated with high rates of morbidity and mortality.

Patients with nonimmunological diseases, secondary immunodeficiencies, nonpharmacological iatrogenic factors, and immunosuppressive drug therapies will be involved in the study.

DETAILED DESCRIPTION:
Severe, up to potentially fatal infections , represent a frequent cause of hospitalization in various clinical settings (pediatric and adult). Any infection of bacterial, viral, mycobacterial, or fungal etiology with a severe course, whether systemic (e.g., sepsis or septic shock, disseminated intravascular coagulation) or focal (e.g., pneumonia, meningitis, encephalitis skin infection) that causes organ damage and/or requires organ-specific or intensive supportive treatment (mechanical ventilation, inotropes, renal replacement treatment) should be considered life-threatening.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent;
* Otherwise healthy patient on admission

Infectious episode:

* life-threatening caused by known or unknown etiologic agent including viruses, bacteria, mycobacteria or mycetes (in case of lack of microbiologic isolate if clinical, laboratory, histopathologic and radiologic data, justify an infectious origin)
* or caused by vaccine strains of attenuated vaccines such as Measles, Mumps, Rubella, Yellow Fever.
* or caused by viruses, bacteria, mycobacteria or mycetes with features suggestive of congenital deficiency of immunity, the clinical pictures below refer to known conditions potentially associated with congenital errors of innate immunity

Viral susceptibility:

* ARDS caused by influenza virus type A, Sars-Cov2
* Life-threatening enterovirus rhomboencephalitis
* Life-threatening infection by VZV, CMV, EBV, Rhinovirus, Respiratory Syncytial Virus
* HSV encephalitis
* Fulminant hepatitis from HAV
* Kaposi's sarcoma from HHV8
* Beta-HPV infections such as: epidermodysplasia verruciformis, mucocutaneous carcinoma,recurrent/diffuse skin warts,, papillomatosis.

Susceptibility to pyogenic bacteria:

* At least one life-threatening infection or two episodes of invasive infectionsin otherwise healthy patients, either systemic (bacteremia) or focal (pneumonia, meningitis, arthritis, osteomyelitis, deep brain/peritoneal/hepatosplenic/muscle abscesses)
* At least two episodes of disseminated or severe staphylococcal muco-cutaneous infections in otherwise healthy patients: decalvant folliculitis, pustules, furunculosis, blepharitis, lymphadenitis, abscesses

Susceptibility to Tropherymawhipplei:

- Whipple's disease

Susceptibility to Mycobacteria:

* Life-threatening , recurrent, or persistent infections with tuberculous or nontuberculous mycobacteria in otherwise healthy patients
* Post-vaccinal BCG-osis from attenuated M. Bovis strain

Susceptibility to mycetes:

* Chronic muco-cutaneous candidiasis Invasive fungal infections of sinuses, lungs, CNS, bones, joints, liver, spleen, and mucocutaneous membranes by Coccidioides, Paracoccidiodes, Cryptococcus, Histoplasma, Pneumocystis, Aspergillus, Talaromyces, Mucormycetes, or Blastomyces
* Invasive candidiasis of brain, eyes, heart, bone, and blood in the absence of central catheters
* Blood dissemination of fungal pathogens (except for candidiasis from central access)
* Persistent positive fungal culture after adequate therapy in terms of drug susceptibility, dosage and duration
* Deep infection with dermatophytes (Microsporum, Epidermophyton, Tricophyton) at dermal and lymph node level
* Infection with rare yeasts (Geotrichum, Kodamaea, Malassezia/Rhodotorula, Saccharomyces, Trichosporon) or rare molds (AureobasidiumChrysosporium, Corynesprora, Exophiala, Geosmithia, Ochroconis, Paecilomyces, Phellinus, Phialophora, Rhizopus, Scopulariopsis)

Other:

-All infectious diseases not included in the list whose natural history differs from that expected for the identified pathogen with regard to severity, recurrence, and persistence of the disease, if the condition is not otherwise explainable by the patient's acquired risk factors.

Exclusion Criteria:

* Patients with nonimmunological diseases, secondary immunodeficiencies, nonpharmacological iatrogenic factors, immunosuppressive drug therapies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Will be enrolled, patients evaluated or admitted, at the O.U. Department of Emergency Pediatrics, Emergency Room and Short and Intensive Observation, the Immunology Outpatient Clinic of the O.U. of Infectious Diseases, the U. O. Anesthesiology and General and Pediatric Resuscitation, of Neonatology and Neonatal Intensive Care, belonging to the IRCCS AOUBO, and the U.O.C. of Pediatric Neuropsychiatry of the IRCCS Institute of Neurological Sciences in Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Identification and Prevalence of cases potentially associated with ECI | through study completion, an average of 1 year
  Identification and calculation of the prevalence of cases potentially associated with ECI (with or without genetic confirmation) among otherwise healthy patients admitted with severe or life-threatening infectious disease

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Zama, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (6):
- Italy (6):
  - IRCCS Istituto delle Scienze Neurologiche, Bologna, Bologna
  - IRCCS Azienda Ospedaliero Universitaria di Bologna UO Pediatria, Bologna, Bologna
  - IRCCS Azienda-Ospedaliero Universitaria di Bologna UO Anestesiologia e Rianimazione generale e pediatrica, Bologna, Bologna
  - IRCCS Azienda-Ospedaliero Universitaria di Bologna UO Malattie Infettive, Bologna, Bologna
  - IRCCS Azienda-Ospedaliero Universitaria di Bologna UO Neonatologia e terapia intensiva neonatale, Bologna, Bologna
  - IRCCS Azienda-Ospedaliero Universitaria di Bologna UO Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve e Intensiva, Bologna, Bologna

IPD SHARING:
Plan to Share IPD: No